CLINICAL TRIAL: NCT06815757
Title: Unveiling Dysphagia in Pediatric Dystonia: Insights From a Cross-Sectional Study
Brief Title: İnvestigating Dysphagia in Pediatric Dystonia
Status: Active, not recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Muserrefe Nur Keles, Assisstant Professor, Gazi University
Other Study IDs: 822426
Record Dates: First submitted 2025-02-01; First posted 2025-02-07 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Dystonia Disorder
Keywords: Dystonia; Pediatric; Dysphagia; DDS
MeSH Terms: conditions — Dystonic Disorders; Dystonia; Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dystonic Children: Children diagnosed with dystonia as the predominant movement disorder

SUMMARY:
Dystonia is a movement disorder involving involuntary, sustained, or intermittent muscle contractions that cause abnormal postures and repetitive movements, worsened by voluntary actions or stress. It is linked to dysfunctions in the basal ganglia, thalamus, and cerebellum, affecting sensorimotor integration. In children, dystonia often coexists with other disorders like spasticity in cerebral palsy, complicating diagnosis and treatment.

Dystonia can be genetic, caused by mutations, or acquired, associated with conditions such as cerebral palsy, perinatal brain injury, and metabolic disorders. A key complication of pediatric dystonia is swallowing dysfunction (oropharyngeal dysphagia), which impairs airway protection and nutrition, increasing the risk of aspiration pneumonia. Studies have shown swallowing impairments across all phases (oral, pharyngeal, and esophageal) in children with dyskinetic cerebral palsy.

However, due to pathophysiological differences between dystonia and cerebral palsy, generalizing findings may lead to inaccuracies. Each dystonia subtype presents unique challenges that affect swallowing function, emphasizing the need for condition-specific assessment and interventions. This study aims to fill the research gap by exploring the clinical features of swallowing dysfunction in children with dystonia, providing insights to improve care and outcomes.

DETAILED DESCRIPTION:
Dystonia is a neurological disorder characterized by involuntary muscle contractions that cause abnormal postures and repetitive movements. These symptoms are often exacerbated by voluntary actions or stress. The condition is linked to dysfunctions in brain regions responsible for motor control, including the basal ganglia, thalamus, and cerebellum, which disrupt sensorimotor integration. In children, dystonia frequently coexists with other neurological disorders, particularly cerebral palsy, making diagnosis and management more complex.

The etiology of dystonia is both genetic and acquired. Genetic forms, though rare, are associated with progressive motor impairments due to mutations in genes. Acquired dystonias are more common and are linked to risk factors like perinatal brain injury, cerebral palsy, and metabolic disorders. Children with dyskinetic cerebral palsy are particularly vulnerable, as their condition shares clinical features with dystonia.

A key complication in pediatric dystonia is oropharyngeal dysphagia, a disorder affecting the ability to swallow. Swallowing requires precise neuromuscular coordination across oral, pharyngeal, and esophageal phases. Disruptions in this process can lead to malnutrition, dehydration, and aspiration pneumonia. Studies on dyskinetic cerebral palsy have highlighted impairments in all phases of swallowing, but due to differences in muscle activation and positioning risks, these findings may not fully apply to children with dystonia.

Each dystonia subtype presents unique clinical challenges. For instance, children with spastic cerebral palsy face high risks of aspiration in a supine position, while children with dystonia may tolerate this position better. Therefore, individualized assessments are essential to ensure accurate diagnosis and treatment.

This study aims to explore the clinical characteristics of swallowing dysfunction in children with dystonia. By investigating how various causes influence its presentation, we seek to develop better diagnostic tools and treatment strategies to improve patient care and quality of life.

ELIGIBILITY:
Inclusion Criteria:

- a confirmed neurological diagnosis, such as cerebral palsy, metabolic disorders, or genetic syndromes, with dystonia as the predominant movement disorder.

Exclusion Criteria:

* encompassed conditions that could interfere with the evaluation process, including active or untreated seizures and acute medical illnesses, such as mouth ulcers, tonsillitis, pharyngitis, or pneumonia.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who were diagnosed predominant movement disorder with dystonia
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-04-17 (Estimated)

PRIMARY OUTCOMES:
Swallowing Disorder Severity | Baseline
  Swallowing disorder severity will be determined using the Dysphagia Disorder Survey (DDS), a validated tool for children aged two years and older. The DDS, which has demonstrated strong internal consistency and validity, includes 15 items divided into two sections: Part 1 assesses related factors such as body mass index, diet, independence, postural control, diet consistency, adaptive utensils, special feeding techniques, and seating alignment, while Part 2 evaluates feeding and swallowing competency, including orienting, food reception, containment, oral transport, chewing, oral-pharyngeal swallowing, post-swallow, and oesophageal swallowing. In line with the developers' recommendations, items 1 and 15 were excluded from the scoring due to weak associations with other items, resulting in total scores ranging from 0 to 34. Higher scores indicated greater swallowing disorder severity.

SECONDARY OUTCOMES:
Aspiration Risk and Swallowing Function Assessment | Baseline
  Aspiration risk will be assessed using the 3-ounce water swallow test. Each child will be asked to drink 3 ounces of water from a cup without interruption while their natural position. If the patient is unable to hold the cup, the clinician assists them. Referral for further assessment will be warranted if the child exhibited coughing, choking, or wet/hoarse vocal quality during or within one minute of completing the test. Performance will be scored as "successful" if no signs of impaired safety were observed and "failed" if any of the criteria were met. In addition, the Pediatric Assessment Tool-10 (PEDI-EAT-10)questionnaire, a parent-proxy tool, will be administered to assess penetration and aspiration risks. This 10-item questionnaire, scored on a 5-point ordinal scale, identified higher risk of unsafe swallowing with increasing scores. A score of ≥4 indicated swallowing dysfunction, and a score of ≥13 indicated a heightened risk of aspiration.

OTHER OUTCOMES:
Assessment of Oral Structure | Baseline
  As part of the oral structure assessment, various observations were made. The presence or absence of open mouth posture and open bite was observed and recorded. Additionally, the presence of tongue thrust and a high-arched palate was assessed.
Assesment of Oral Hygiene | Baseline
  Oral hygiene was evaluated by counting the number of missing, filled, or decayed teeth. The presence of halitosis (bad breath) and daily tooth brushing habits were also recorded. Tooth brushing was noted as "present" if it occurred at least once daily.

CONTACTS AND LOCATIONS:
Overall Officials: Muserref Keles, PhD, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided